CLINICAL TRIAL: NCT03659669
Title: Post Marketing Observational Study to Describe the Effectiveness and Safety of Venetoclax Treatment in Chronic Lymphocytic Leukemia (CLL) Patients in Routine Clinical Practice
Brief Title: A Study to Describe the Effectiveness and Safety of Venetoclax Treatment in Chronic Lymphocytic Leukemia (CLL) Patients in Routine Clinical Practice
Acronym: REVEAL
Status: Suspended | Type: Observational
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P19-287
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: Chronic Lymphocytic Leukemia; Cancer; venetoclax; observation
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Chronic Lymphocytic Leukemia (CLL): Patients with diagnosed CLL and eligible to venetoclax as per label.

SUMMARY:
This study will evaluate effectiveness and safety in routine clinical practice in participants starting venetoclax treatment for Chronic Lymphocytic Leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

* Participants with diagnosed Chronic Lymphocytic Leukemia (CLL) and eligible for venetoclax as per label.
* Participants for whom the physician has decided to initiate CLL treatment with venetoclax.
* Participants who have been informed verbally and in writing about this study, and who do not object to their data being processed or subjected to data quality control.

Exclusion Criteria:

- Participants currently participating (or previously participated) in an interventional clinical trial within 30 days prior to venetoclax treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with diagnosed CLL and receiving venetoclax as per label.
Sampling Method: Non-Probability Sample
Enrollment: 272 (Estimated)
Dates: Start 2019-02-10 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 12 months
  ORR to treatment is defined as the proportion of patients with complete response (CR), Complete Response with incomplete bone marrow recovery (CRi), nodular Partial Response (nPR) and partial response (PR), according to physician's assessment.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to approximately 24 months
  ORR to treatment is defined as the proportion of patients with complete response (CR), Complete Response with incomplete bone marrow recovery (CRi), nodular Partial Response (nPR) or partial response (PR), according to physician's assessment.
Complete Response (CR) Rate | Up to approximately 24 months
  CR is defined as the proportion of participants with either CR and CRi, according to physician's assessment.
Time to Response (TTR) | Up to approximately 24 months
  TTR is defined by the time between the date of the first venetoclax intake and the date of the first assessment having documented the response among complete response, complete response with incomplete bone marrow recovery, nodular partial response, and partial response.
Time to Best Response to Treatment | Up to approximately 24 months
  The time to best response to treatment is defined by the time between the date of the first venetoclax intake and the date of the assessment having documented the best response among CR, CRi, nPR, and PR.
Overall Survival (OS) | Up to approximately 48 months
  Overall survival (OS) is defined as the time from the date of first venetoclax intake to the date of death from any cause.
Time To Progression (TTP) | Up to approximately 48 months
  The Time To Progression (TTP) is defined as the time from the date of first venetoclax intake to the date of the first documented disease progression.
Progression-Free Survival (PFS) | Up to approximately 48 months
  PFS is defined as the time from the date of first venetoclax intake to the date of the first documented disease progression or death from any cause.
Time To Next Treatment | Up to approximately 48 months
  Time to next treatment is defined as the time between the date of the first venetoclax intake and the date of the first next treatment intake after venetoclax discontinuation.
Duration of Response (DOR) | Up to approximately 48 months
  DOR is calculated in the sub-population of patients experiencing treatment response (complete response, complete response with incomplete bone marrow recovery, nodular partial response or partial response) from the date when response is first met to the date of first following documented progression.
PFS after Disease Progression Following Venetoclax Treatment | Up to approximately 48 months
  PFS following venetoclax treatment is defined as the time from the date of first next CLL treatment intake to the date of the following documented progression or death from any cause.
Best Response under Next CLL Treatment | Up to approximately 48 months
  The best response under next CLL treatment is calculated in the sub-population of participants having a next CLL treatment after venetoclax discontinuation.
Minimal Residual Disease | Up to approximately 24 months
  The proportion of participants with assessment of the minimal residual disease under venetoclax treatment (assessed by flow cytometry or Polymerase Chain Reaction).
Change in Score of EuroQol 5 Dimensions (EQ-5D-5L) | Up to approximately 24 months
  The EQ-5D-5L has five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. These dimensions are measured on a five-level scale: no problems, slight problems, moderate problems, severe problems, and extreme problems. The scores for the 5 dimensions are used to compute a single utility index score ranging from zero (0.0) to 1 (1.0) representing the general health status of the individual. The EQ-5D-5L also contains a visual analog scale (VAS) to assess the subject's overall health.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (13):
- Israel (13):
  - Soroka University Medical Center /ID# 207897, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 207900, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 206962, Tel Aviv, Tel Aviv
  - HaEmek Medical Center /ID# 210900, Afula
  - Rambam Health Care Campus /ID# 210320, Haifa
  - Bnai Zion Medical Center /ID# 206963, Haifa
  - Shaare Zedek Medical Center /ID# 207896, Jerusalem
  - Hadassah /ID# 207898, Jerusalem
  - Meir Medical Center /ID# 215466, Kfar Saba
  - Galilee Medical Center /ID# 207899, Nahariya
  - Rabin Medical Center /ID# 206961, Petah Tikva
  - Kaplan Medical Center /ID# 207902, Rehovot
  - Ziv Medical Center /ID# 215462, Safed

IPD SHARING:
Plan to Share IPD: Undecided